CLINICAL TRIAL: NCT00300963
Title: A Multicenter, Double-Blind, Double-Dummy, Placebo-Controlled, Randomized, Parallel Group Evaluation of the Efficacy and Safety of a Fixed-Dose of Talnetant Versus Placebo Versus Risperidone in Subjects With Schizophrenia
Brief Title: Effect Of Talnetant Versus Risperidone Versus Placebo On Psychotic Symptoms In Schizophrenic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 223412/093
Record Dates: First submitted 2006-03-07; First posted 2006-03-10 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: psychosis; cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — SB 223412

INTERVENTIONS:
Drug: Talnetant

SUMMARY:
The purpose of this study is to test the safety and effectiveness of talnetant vs. risperidone vs. placebo in reducing positive and negative symptoms in acutely psychotic schizophrenia patients.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have schizophrenia which is not secondary to another medical condition or substance abuse.
* Require inpatient hospitalization.
* Women may enroll only if they are not of child-bearing potential OR are on a protocol-approved birth control method.

Exclusion criteria:

* Subject is in their first episode of schizophrenia.
* Subject has other psychotic disorders or bipolar disorder.
* Subject has schizophrenia symptoms from taking another medicine or drug of abuse, or due to a general medical condition.
* Subject has a recent history of substance dependence, or tests positive for illicit drug.
* Subject has an unstable medical disorder, or any significant medical disorder including autistic disorder, organic brain disease, liver dysfunction, epilepsy or seizures, or is at increased risk of developing cerebrovascular problems like stroke.
* Subject has any significant abnormalities in any of the screening tests (ECGs, labs, physical examinations, etc.).
* Subject poses a current serious suicidal or homicidal risk.
* Subject has a positive pregnancy test, or is lactating or planning to become pregnant within one month of the study.
* Subject has recently or is currently participating in another clinical study.
* Subject is stabilized on their current schizophrenia treatment.
* Subject needs to take any of the medicines not permitted in the study, or has recently had ECT (electroconvulsive therapy) or TMS (transcranial magnetic stimulation).
* Subject was non-responsive to two or more adequate trials of antipsychotic treatments over the past 2 years.
* Subject has had an allergic or significant reaction to any of the study drugs, or can't take risperidone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275
Dates: Start 2004-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is change in the Positive and Negative Syndrome Scale (PANSS) at Week 6 compared to baseline values.

SECONDARY OUTCOMES:
The secondary measures assess both efficacy (cognition, depression) as well as a variety of safety/tolerability endpoints (adverse events, motor function, laboratory measures).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (20):
- United States (20):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Pico Rivera, California
  - GSK Investigational Site, Rosemead, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Richmond, Virginia